CLINICAL TRIAL: NCT00451620
Title: Effect of GlucoNorm vs Glyburide on Post-Prandial Hyperglycemia in Elderly Subjects With Type 2 Diabetes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Novo Nordisk A/S (Industry)
Responsible Party: Principal Investigator, Graydon Meneilly, Principal Investigator, University of British Columbia
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: H02-70584; H02-70584
Record Dates: First submitted 2007-03-21; First posted 2007-03-23 (Estimated); Last update posted 2018-01-18 (Actual); Status verified 2018-01

CONDITIONS: Type 2 Diabetes
Keywords: Type 2 diabetes; Hypoglycemia; Oral hypoglycemic agents; Insulin levels
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Hypoglycemia | interventions — Glyburide; repaglinide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 2. (Experimental): GlucoNorm
  Interventions: Drug: GlucoNorm
- 1. (Experimental): Glyburide
  Interventions: Drug: glyburide

INTERVENTIONS:
Drug: glyburide — Subjects will undergo 2 Standard Meal Tests with Ensure 325 ml separated by 15 - 30 days. Group 1 will receive GlucoNorm 1 mg during the 1st Standard Meal Test and Glyburide 2.5 mg during the 2nd Standard Meal Test. Group 2 will receive Glyburide 2.5 mg during the 1st Standard Meal Test and GlucoNorm 1mg during the 2nd Standard Meal Test.
  Arms: 1.
Drug: GlucoNorm — Subjects will undergo 2 Standard Meal Tests with Ensure 325 ml separated by 15 - 30 days. Group 1 will receive GlucoNorm 1 mg during the 1st Standard Meal Test and Glyburide 2.5 mg during the 2nd Standard Meal Test. Group 2 will receive Glyburide 2.5 mg during the 1st Standard Meal Test and GlucoNorm 1mg during the 2nd Standard Meal Test.
  Arms: 2.

SUMMARY:
The results from the DECODE Study have shown that postprandial (1 - 2 hours after a meal) hyperglycemia (elevated blood sugar) is more common in elderly people with diabetes than younger people with diabetes and is the best predictor of the development of complications. The DECODE Study involved 6941 people who already had diabetes and 702 who did not have diabetes. Diabetes is diagnosed when the blood sugar 1st thing in the morning is over 7.0 mmol/L. The DECODE Study showed that people at risk for diabetes can have a normal blood sugar 1st thing in the morning but have a high blood sugar 2 hours after a meal and that these people are at risk for developing heart disease and other complications of diabetes. These people would not be identified as at risk if only a fasting blood sugar is done. Studies in younger people with diabetes have shown that after a meal, insulin levels are more like a person without diabetes and glucose (blood sugar) levels are lower with GlucoNorm than with Glyburide. There is no data available that demonstrates this in elderly people with type 2 diabetes.

You have been invited to participate in this study because you have type 2 diabetes controlled by diet and/or exercise or metformin only and are over 65 years of age.

The purpose of this study is to determine whether GlucoNorm has a greater effect than Glyburide on insulin levels and glucose (blood sugar) levels after a meal in elderly people with type 2 diabetes who control their diabetes with diet and exercise.

DETAILED DESCRIPTION:
The results from the DECODE Study have shown that postprandial hyperglycemia is more common in elderly people with diabetes than younger people and is the best predictor of mortality and morbidity. Studies in younger people with diabetes have shown that in response to a meal, insulin profiles are more physiologic and glucose levels are lower with GlucoNorm than with Glyburide. There is no data available that demonstrates this in elderly people with type 2 diabetes.

This is a randomized, open-label, cross-over study. Subjects will undergo 2 Standard Meal Tests with Ensure 325 ml separated by 15 - 30 days. Group 1 will receive GlucoNorm 1 mg during the 1st Standard Meal Test and Glyburide 2.5 mg during the 2nd Standard Meal Test. Group 2 will receive Glyburide 2.5 mg during the 1st Standard Meal Test and GlucoNorm 1mg during the 2nd Standard Meal Test.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes > 3 months duration
* Male or female
* Over 65 years of age
* Diet controlled only
* HgbA1C < 8.5%

Exclusion Criteria:

* Treatment with oral hypoglycemic agents or insulin or the likelihood of requiring treatment with these during the study.
* Anemia - hgb below 130 g/L (males) and below 120 g/L (females).
* Taking medications that known to interfere with glucose metabolism eg systemic corticosteriods, non-selective beta blockers.
* Known or suspected allergy to glyburide, sulfa drugs or GlucoNorm impaired liver function, as shown by but not limited to AST and/or ALT > 2x the upper limit of normal.
* Impaired renal function, as shown by but not limited to serum creatinine > 133 µmol/L (males) or 124 µmol/L (females).
* Participated in another clinical trial within the past 30 days.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 30 (Actual)
Dates: Start 2003-11; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
The objective of this study is to determine whether GlucoNorm has a greater effect than Glyburide on insulin levels and postprandial glucose levels in elderly people with type 2 diabetes who are diet controlled. | 2 hours

CONTACTS AND LOCATIONS:
Overall Officials: Graydon Meneilly, MD, Principal Investigator — University of British Columbia
Locations (1):
- University of British Columbia, Vancouver, British Columbia, Canada